CLINICAL TRIAL: NCT02205008
Title: Prospective Randomized Multicenter Phase III Trial of Intraperitoneal Chemotherapy and Systemic Chemotherapy Versus Systemic Chemotherapy After Curative Resection of Serosa-positive Gastric Cancer
Brief Title: Intraperitoneal Chemotherapy and Systemic Chemotherapy Versus Systemic Chemotherapy After Curative Resection of Serosa-positive Gastric Cancer
Acronym: EPIC-GC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kyungpook National University Hospital (Other)
Collaborators: National Cancer Center, Korea (Other Government); Keimyung University Dongsan Medical Center (Other); Yeungnam University Hospital (Other); Daegu Catholic University Medical Center (Other); Chonnam National University Hospital (Other); Dong-A University Hospital (Other); Severance Hospital (Other); Korea Cancer Center Hospital (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Hanyang University (Other)
Responsible Party: Principal Investigator, Wansik Yu, professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPIC-GC; KNUMCGCC-001 (Other: KNUMC)
Record Dates: First submitted 2014-07-26; First posted 2014-07-31 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Advanced Gastric Cancer With Serosal Invasion
Keywords: advanced gastric cancer; serosal invasion; peritoneal recurrence; intraperitoneal chemotherapy
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Active Comparator): curative resection of the stomach with D2 plus intraperitoneal chemotherapy plus adjuvant systemic chemotherapy with S-1
  Interventions: Procedure: surgery; Drug: adjuvant systemic chemotherapy; Drug: Early postoperative intraperitoneal chemothgerapy
- Arm B (Placebo Comparator): curative resection of the stomach with D2 plus adjuvant systemic chemotherapy with S-1
  Interventions: Procedure: surgery; Drug: adjuvant systemic chemotherapy

INTERVENTIONS:
Procedure: surgery — Total or subtotal gastrectomy with D2
Drug: adjuvant systemic chemotherapy — adjuvant systemic chemotherapy with S-1 (<1.25m2:40mg, 1.25-1.5m2:50mg, >1.5m2:60mg, bid)
Drug: Early postoperative intraperitoneal chemothgerapy — operation day: 0.9％ saline solution 1L plus mitomycin C 10 mg/m2
  1 - 4 postoprative day: 0.9％ saline solution 1L plus 5-FU 700 mg/m2 plus sodium bicarbonate 50 mEq
  Arms: Arm A

SUMMARY:
Intraperitoneal chemotherapy as an adjuvant treatment modality is designed to eradicate intraperitoneal free tumor cells that can be a source of peritoneal carcinomatosis. Although we have not reached unanimous consensus, favorable reports on the outcome of intraperitoneal chemotherapy have been published.

In this study, we review the clinicopathological characteristics of patients and effects of early postoperative intraperitoneal chemotherapy (EPIC) on overall and gastric cancer-specific survival and patterns of recurrence of gastric cancer patients with macroscopic serosal invasion.

The aim of this study is to evaluate the impact of intraperitoneal chemotherapy on overall and disease free survival of advanced gastric cancer patients with serosal invasion after potentially curative surgery.

ELIGIBILITY:
Inclusion Criteria:

1. histologically proven adenocarcinoma of the stomach
2. preoperative suspicion of serosal invasion on the radiological examination
3. candidate for curative resection of the stomach with D2
4. age from 19 to 70 year old
5. Eastern Cooperative Oncology Group Performance status :0, 1, or 2
6. absolute neutrophil count≥1,500/microliter, hemoglobin≥9.0g/dL, and platelet≥100,000/microliter
7. serum Creatinine<1.5mg/dL
8. total bilirubin <2 x upper normal limit, transaminase<3 x upper normal limit
9. patients without previous administration of chemotherapeutic agent
10. patients who agreed and signed to the informed consent form

Exclusion Criteria:

1. malignancy of the stomach except for adenocarcinoma
2. history of hypersensitivity to 5-fluorouracil or mitomycin
3. concomitant infectious disease
4. active hepatitis or chronic liver disease
5. history of psychotic disorders
6. patients with disorders in the central nervous system
7. history of other malignancy within 5 years
8. history of clinically significant heart disease (congestive heart failure, symptomatic coronary artery disease, symptomatic arrhythmia, myocardial infarction)
9. patients with increased bleeding tendency
10. pregnant or lactating female patients
11. patient who did not agreed and signed to the informed consent form

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2012-10; Primary Completion 2015-12 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
relapsed free survival | postoperative 3 years
  during regular follow-up with blood test, radiologic, endoscopic surveillance patients with recurrence will be detected and recorded

SECONDARY OUTCOMES:
overall survival | postoperative 5 years
  during regular follow-up with blood test, radiologic, endoscopic surveillance patients with recurrence will be detected and recorded

OTHER OUTCOMES:
surgery and intraperitoneal chemotherapy-related morbidity and mortality | postoperative 30days
  In hospital complication related to surgery or intraperitoneal chemotherapy will be recored and analyzed to evaluate the safety of intraperitoneal chemotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Wansik Yu, MD. PhD, Principal Investigator — Kyungpook National University Medical Center
Locations (1):
- Kyungpook National University Medical Center Gastric Cancer Center, Daegu, South Korea

REFERENCES:
- [Background] 1. Maruyama K, Okabayashi K, Kinoshita T. Progress in gastric cancer surgery in Japan and its limits of radicality. World J Surg 1987;11:418-425. 2. Lee JL, Kang HJ, Kang YK, et al. Phase I/II study of 3-week combination of S-1 and cisplatin chemotherapy for metastatic or recurent gastric cancer. Cancer Chemother Pharmacol 2007 (E-pub). 3. Schoffski P. The modulated oral fluoropyrimidine prodrug S-1, and its use in gastrointestinal cancer and other solid tumors. Anticancer Drug 2004;15:85-106. 4. Sugimachi K, Maehara Y, Horikoshi N et al. An early phase II study of oral S-1, a newly developed 5-fluorouracil derivative for advanced and recurrent gastrointestinal cancers. Oncology 1999;57:202-210. 5. Koizumi W, Kurihara M, Nakajo S et al. Phase II study of S-1, a novel oral derivative of 5-fluorouracil, in advanced gastric cancer. Oncology 2000;58:191-197. 6. Sakata Y, Ohtsu A, Horikoshi N et al. Late phase II study of novel oral fluoropyrimidine anticancer drugs S-1 (1 M tegafur-0.4 M gimestat-1 M otastat potassium) in advanced gastric cancer patients. Eur J Cancer 1998;34:1715-1720. 7. Nagashima F, Ohtsu A, Yoshida S et al. Japanese nationwide postmarketing survey of S-1 in patients with advanced gastric cancer. Gastric Cancer 2005;8:6-11. 8. Chollet P, Schoffski P, Weigang-Kohler K et al. Phase II trial with S-1 in chemotherapy-naïve patients with gastric cancer. A trial performed by the EORTC early clinical studies group (ECGC). Eur J Cancer 2003;39:1264-1270. 9. Ilson D. Just when you thought the fluorouracil debate was over: S-1 and gastric cancer. J Clin Oncol 2005;23:6826-6828. 10. Hoff PM, Saad ED, Ajani JA et al. Phase I study with pharmacokinetics of S-1, an oral daily schedule for 28 days in patients with solid tumors. Clin Cancer Res 2003;9:134-142. 11. Simon R. Optimal two-stage design for phase II clinical trials. Controlled Clin Trials 1989;10:1-10.